CLINICAL TRIAL: NCT03796221
Title: Integrating Parenting Interventions Into Pediatric Obesity Care
Brief Title: Parenting Intervention for Pediatric Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Health System (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Thao-Ly Phan, Associate Professor of Pediatrics, Nemours Children's Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23HD083439 (NIH); K23HD083439 (NIH)
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Childhood Obesity; Parenting
Keywords: Childhood obesity; Parenting intervention; Video intervention; Healthcare delivery
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Will receive standard pediatric obesity treatment
  Interventions: Behavioral: Standard pediatric obesity treatment
- Intervention Group (Experimental): Will receive standard pediatric obesity treatment and parenting videos
  Interventions: Behavioral: Parenting videos; Behavioral: Standard pediatric obesity treatment

INTERVENTIONS:
Behavioral: Parenting videos — Brief online videos, featuring families of children with obesity of diverse backgrounds, to provide education on parenting skills and motivate families to adopt healthy lifestyle behaviors as a family. Videos will be delivered monthly for three months in between pediatric obesity clinic visits.
  Arms: Intervention Group
Behavioral: Standard pediatric obesity treatment — Standard treatment in a hospital-based pediatric obesity clinic with a team of medical providers, dietitians, exercise specialists, and behavioral health specialists. Treatment includes management of obesity-related medical conditions, nutrition education, physical activity counseling, and discussion of behavioral strategies such as goal-setting and self-monitoring, with elements of motivational interviewing used to encourage behavior change and adoption of healthy lifestyle behaviors by the entire family.

SUMMARY:
The purpose of this study is to see if educational videos about how to help children develop healthy behaviors, paired with treatment in a pediatric obesity clinic, can increase caregiver confidence and improve child behaviors and weight. Caregivers of children between the ages of 4 and 11 years old who are new patients to a pediatric obesity clinic will be invited to take part in the study. All families will receive the standard treatment provided in the pediatric obesity clinic. Half of the caregivers will be assigned to also watch a few educational videos every month for 3 months in between clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Legal guardian of a new patient to the Nemours pediatric obesity clinic
* Child with body mass index (BMI) greater than the 95th percentile for age and sex
* Child 4-11 years of age

Exclusion Criteria:

* Not proficient in English or Spanish
* Not able to access the internet on any type of device
* Child has a genetic syndrome or primary endocrine disorder associated with obesity
* Child is taking a medication known to impact weight

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
Change in child weight status | 6 months
  Change in child BMI-z score
Change in child weight status | 6 months
  Change in child BMI percentile (referenced to the 95th percentile)
Change in caregiver confidence managing child lifestyle behaviors | 6 months
  Change in Lifestyle Behavior Checklist Confidence score
Change in child lifestyle behaviors | 6 months
  Change in Lifestyle Behavior Checklist Problem score

SECONDARY OUTCOMES:
Discussion of parenting topics during visits to the pediatric obesity clinic | 1 month, 2 months, 3 months, 6 months
  Discussion helpfulness ratings at each visit
Change in child weight status | 3 months
  Change in child BMI-z score
Change in child weight status | 3 months
  Change in child BMI percentile (referenced to the 95th percentile)
Change in caregiver confidence managing child lifestyle behaviors | 3 months
  Change in Lifestyle Behavior Checklist Confidence score
Change in child lifestyle behaviors | 3 months
  Change in Lifestyle Behavior Checklist Problem score

CONTACTS AND LOCATIONS:
Overall Officials: Thao-Ly T Phan, MD MPH, Principal Investigator — Nemours Children's Health System
Locations (1):
- Nemours Alfred I. duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No